CLINICAL TRIAL: NCT04365296
Title: Aerobic Versus Resistance Exercises on Liver Enzymes Following Burn Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Gamal Fawzy El-Sayed (Other)
Responsible Party: Sponsor-Investigator, Aya Gamal Fawzy El-Sayed, Assistant lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002230
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic group (Experimental): This group will include 30 burned patients who will receive aerobic exercises 8 weeks (3times/week) in form of treadmill exercise in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment (medications as cataflam, alphintern, zinetac and hemacaps and wound dressings).
  Interventions: Other: Experimental
- Resistance group (Experimental): This group will include 30 burned patients who will receive resistance exercises 8 weeks (3times/week) by using dumbbells and sand bags in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment (medications as cataflam, alphintern, zinetac and hemacaps and wound dressings).
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — The purpose of the study is to evaluate which is more effective aerobic or resistance exercises in reducing plasma liver enzymes level (AST and ALT) post burn. Subjects and Methods: Sixty burned patients with burned body surface area about 30% to 50% will participate in this study. Their ages will be ranged from 20-45 years. They will be selected from Orabi Hospital and will be divided randomly into two equal groups.

SUMMARY:
1. Subjects:

   Sixty patients suffering from partial thickness burn with burned body surface area (BBSA) about 30% to 50% will be randomly divided into two equal groups each one has 30 patients.
2. Equipment and tools:

2.1. Measurement equipment: Spectrophotometer device. 2.2. Therapeutic equipment and tools: Treadmill device for aerobic exercises and dumbbells and sand bags for resistance exercises.

DETAILED DESCRIPTION:
Sixty patients who have partial thickness burn with burned body surface area (BBSA) about 30% to 50% will participate in this study after their release from intensive care unit. Their ages will be ranged from 20 to 45 years. The participants will be selected from Orabi hospital and randomly distributed into two equal groups. In this study the patients will be randomly assigned into two equal groups (30 patients for each group):

1.1(a) Group A (Aerobic exercise group): This group includes 30 burned patients who will receive aerobic exercises 8 weeks (3times/week) in form of (treadmill device) in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment.

1.1(b) Group B (Resistance exercise group): This group includes 30 burned patients who will receive resistance exercises 8 weeks (3times/week) by using dumbbells and sand bags in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment.

3.1-Measurement procedures:

* Serum blood draws will be taken by certified technicians with the participant in a seated position.
* Spectrophotometry is the measurable analysis technique using the electromagnetic spectra. It deals with the ranges of wavelengths such as near ultraviolet, near infrared and visible light. A device called a spectrophotometer is used to measure the absorbance or transmittance through a liquid sample. The spectrophotometer takes a measurement at a specific wavelength and it is possible to choose any wavelength in the spectrophotometers register as the double beam sends a beam through a blank reference sample and one through the sample to be measured (Nilsson, 2010).

3.2-Therapeutic procedures: 3.2.a- Treadmill device for aerobic exercise: During the 8-week intervention period, an aerobic training (AT) program of submaximal intensity will include a 45-minute session three times a week (135 min/week) under the supervision of the researcher. Aerobic exercise will consist of three phases: warm-up, training and cool down. At the beginning of exercise session, subjects will have a ten-minute warm-up. The warmup protocol will be slowly running on treadmill. Then, the warm-up phase will be followed by the training phase. At baseline, the training phase will be commenced with two 15-minute running on treadmill at 60% of their maximal heart rate (MHR) in the first week and increased to two 15-minute running on treadmill at 75% MHR per week by the final week of training. By the end of exercise session, subjects will have a five-minute cool down. The cool down protocol will be slowly running on treadmill (Khalighfard et al., 2011).

Maximum heart rate will be calculated using the formula: (HRMax =220- age) (Chaudhary et al., 2010).

3.2.b- Dumbbells and sand bags for resistance exercise: Resistance training will be performed during 8-weeks with thrice weekly sessions on nonconsecutive days. The program will consist of seven exercises: triceps press, biceps curl, lat pull down, calf raise, leg press, leg extension and sit-ups using dumbbells and sand bags. Each session will last approximately 45 minutes and consist of a 5-minute warm-up with stretching following by resistance exercise that will be done as a cir¬cuit, ending with 5-minute cool down. The 1 repetition maximum (1RM) is measured at baseline and follow¬ing the intervention. Initially, participants will do two circuits using 50% of their 1RM and repeat them 10 times for the first and second weeks, progressing to two circuits, using 60% of their 1RM and repeat 10 times for the third and fourth weeks. In fifth and sixth weeks, participants will do three circuits using 60% of their 1RM and repeat 10 times. In the last two weeks, patients will do three circuits using 70% of their 1RM and repeat 10 times. A 90-second rest will be allowed between sets of exercises (Hallsworth et al., 2011).

ELIGIBILITY:
Inclusion Criteria:

* -The subject selection will be according to the following criteria:
* Age range between 20-45 years.
* Male and female patients will participate in the study.
* All patients have burn with BBSA about 30% to 50%.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Cardiac diseases.
* Burn of sole of foot.
* Exposed hand or foot tendons.
* Lower limb amputation.
* History of liver diseases.
* Body mass index (BMI=kg/cm2)<30%.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Measures of AST and ALT Liver enzymes post treatment | 2 months
  Measures of AST and ALT Liver enzymes post 8 weeks of treatment for 10 patients of Aerobic group and 10 patients of resistance group.

CONTACTS AND LOCATIONS:
Overall Officials: A M Abd El Baky, Prof.DR, Study Chair — Cairo University
Locations (1):
- Orabi Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No